CLINICAL TRIAL: NCT07177924
Title: Effectiveness, Safety and Learning Curve of Monarch Robotic Assisted Bronchoscopy for Lung Nodule ICG Dye Marking Before VATS Sublobectomy
Brief Title: Monarch Robotic Bronchoscopy for Lung Nodule ICG Dye Marking Before VATS
Acronym: REALM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025YJZ92
Record Dates: First submitted 2025-08-27; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Small Pulmonary Nodules; Pulmonary Nodule Localization; Lung Cancer (Suspected or Confirmed); Video-assisted Thoracoscopic Surgery (VATS)
Keywords: Robotic Assisted Bronchoscopy; Monarch Platform; Lung Nodule Localization; Video-Assisted Thoracoscopic Surgery (VATS); Pulmonary Nodules; Lung Cancer Surgery
MeSH Terms: conditions — Lung Neoplasms; Multiple Pulmonary Nodules

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, single-arm interventional study in which all enrolled patients with small pulmonary nodules difficult to localize during VATS will undergo preoperative indocyanine green (ICG) mixed with iodinated contrast dye marking under Monarch Robotic Assisted Bronchoscopy (RAB) with Cone-Beam CT (CBCT) guidance, immediately followed by VATS sublobectomy in the same operative session. The localization procedure is performed by a single surgeon without prior RAB localization experience to evaluate the learning curve.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Monarch RAB + CBCT-guided ICG Localization + VATS Sublobectomy (Experimental): All participants will undergo preoperative localization of small pulmonary nodules using indocyanine green (ICG) mixed with iodinated contrast agent under Monarch Robotic Assisted Bronchoscopy (RAB) with Cone-Beam CT (CBCT) guidance, performed by a single surgeon without prior RAB localization experience. Immediately after localization, patients will undergo video-assisted thoracoscopic surgery (VATS) sublobectomy (wedge resection or segmentectomy).
  Interventions: Procedure: Monarch RAB with CBCT-guided ICG Dye Marking

INTERVENTIONS:
Procedure: Monarch RAB with CBCT-guided ICG Dye Marking — Under general anesthesia, the Monarch RAB platform is used to navigate to the target bronchus. With CBCT confirmation, 0.25 ml of ICG (0.2 mg/ml) mixed with 0.25 ml iodinated contrast is injected within 1 cm of the nodule. The dye marking is identified intraoperatively with near-infrared light to guide VATS sublobectomy.

SUMMARY:
This is a single-center, prospective, single-arm clinical study conducted at Beijing Cancer Hospital to evaluate the effectiveness, safety, and learning curve of preoperative indocyanine green (ICG) dye marking mixed with iodinated contrast agent under Monarch Robotic Assisted Bronchoscopy (RAB) with Cone-Beam CT (CBCT) for small pulmonary nodules that are difficult to locate during video-assisted thoracic surgery (VATS) sublobectomy. Eligible patients will undergo RAB localization immediately followed by VATS in the same operative session. The primary endpoints include the success rate of localization, effective localization, and VATS sublobar resection. Secondary endpoints include navigation success rate, operation times, reaching depth, complication rates, and health economic outcomes. The learning curve will be analyzed using the cumulative sum (CUSUM) method. A total of 50 patients will be enrolled and followed up for 14 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Clinically indicated sub-lobar resection
* Tolerates general anesthesia
* Single/multiple small nodules <20 mm in peripheral lung field
* Nodules difficult to locate intraoperatively by inspection/palpation

Exclusion Criteria:

* Contraindications to bronchoscopy/anesthesia
* Coagulopathy or bleeding tendency
* Implanted devices interfering with navigation
* Allergy to ICG or iodinated contrast
* Pregnant/lactating women
* Intraoperative findings not suitable for procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of localization procedure | Periprocedural( localization procedure)
  Calculated as (number of successful localization procedures ÷ total localization procedures) × 100%. Success is defined as ICG dye successfully injected at planned target site as confirmed by CBCT. Unit of Measure: participants (%).
Success rate of effective localization | Perioperative (during VATS)
  Calculated as [(number of successful localization procedures - number unrecognized in operative field) ÷ total localization procedures] × 100%. Effective localization is defined as visible ICG staining on pleura during VATS. Unit of Measure: participants (%).
Success rate of VATS sub-lobar resection | Perioperative (during VATS)
  Calculated as (number of successful VATS resections ÷ total localization procedures) × 100%. Successful VATS resection is defined as resection containing the complete lesion and the dye together. Unit of Measure: participants (%).

SECONDARY OUTCOMES:
Learning curve for localization | Through study completion, up to 8 months
  Number of cases required for surgeon to achieve proficiency using cumulative sum (CUSUM) method based on OT1 and localization success rate.Unit of Measure: case number.
Bronchoscopy-related complication rate | From end of bronchoscopy through Postoperative Day 14.
  Incidence of pneumothorax, bleeding, and respiratory failure related to bronchoscopy, graded according to CTCAE. participants (%).
Health economic outcomes | During index hospitalization
  Includes postoperative hospital stay, total hospitalization cost, complication treatment cost, anesthesia cost, and localization procedure cost. Unit of Measure: CNY.

CONTACTS AND LOCATIONS:
Overall Officials: Shaohua Ma, Principal Investigator — Peking University Cancer Hospital & Institute, Beijing 100142, China

IPD SHARING:
Plan to Share IPD: No